CLINICAL TRIAL: NCT05475197
Title: Evaluation of the Acute Effect of Kinesio Taping on Structures at the Wrist Level by Ultrasonography in Patients With Carpal Tunnel Syndrome
Brief Title: Evaluation of the Acute Effect of Kinesio Taping by Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Orhan Güvener, Assistant of Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEUTF-FTR-GUVENER-001
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome,; Ultrasound; Kinesio taping
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping Type 1 (Experimental): For the first group; While the wrist is 30° extension, the forearm is supinated and the elbow is extended, the distance between the 1st metacarpal joint and the medial epicondyles of the patient up to 5 cm below the median epicondyle will be measured. Two strips with width of 2.5 cm will be prepared. For the median nerve, the first band will be adhered along the nerve trachea by stretching of moderate intensity (50%) from the 2nd and 3rd metacarpophalangeal joint to 5 cm below the medial epicondyle.
  The second strip will be applied without stretching to a distance of 5 cm under the medial epicondyle from the 4th and 5th metacarpophalangeal joint. In addition, a strip half the length of the wrist circumference will be adhered to the volar face of the wrist by applying tension to the middle 1/3 of it, without applying tension to both ends.
  Interventions: Device: Kinesio taping
- Kinesio taping Type 2 (Experimental): For the second group; While the elbow is in full extension and the wrist in the extension and supination position, the distal two free ends of the tape will be adhered to the thenar and hypothenar regions without stretching. The middle 1/3 of the X-shaped tape will be adhered to the forearm volar face by applying moderate stretching.The first half of the two proximal free ends will have adhered to the medial and lateral epicondyle with little or no stretching, and the last half without any stretching.
  The I-shaped tape will be adhered to the radial region of the wrist with the elbow in full extension, the wrist in a neutral position, and the palm closed. The middle of the tape will be stretched lightly and moderately, and the last 1/3 of it will be adhered to the ulnar part of the wrist without stretching. Kinesio taping will be applied to both groups once.
  Interventions: Device: Kinesio taping

INTERVENTIONS:
Device: Kinesio taping — We planned to perform two different taping applications to evaluate the acute effect of kinesio taping application on the carpal tunnels of individuals with carpal tunnel syndrome.

SUMMARY:
The design of our study is a randomized, controlled, double-blind study. It is planned to be completed in twenty-four weeks with 34 participants. The main purpose of this study is to examine and compare the acute effects of two different kinesio tape applications on the carpal tunnel in patients with carpal tunnel syndrome by ultrasonographic method.

DETAILED DESCRIPTION:
Methodology of the Study:

This study will make on 15.09.2022 and within 15.01.2023 in the Department of Physical Medicine and Rehabilitation of Mersin University Faculty of Medicine Hospital. Patients who have been diagnosed with carpal tunnel syndrome and whose treatment is planned and who meet the inclusion and exclusion criteria will participate.

Anthropometric measurements:

On the day of arrival for the test, Dr. Figen Dağ (PhD, PT) will measure their height and weight and calculate their body mass index within the scope of anthropometric measurements. The height measurement will be measured by a height meter fixed to the wall. For this, volunteers will be asked to take off their shoes, stand upright and face the other side. BMI values will be calculated by dividing body weights by the square of height (kg/m2). With the bioelectric impedance method (Tanita BC-418 MA, Tanita Corporation, Tokyo, Japan), the body composition (lean body mass, fat mass, fat percentage, etc.) of all individuals will be determined. For this measurement, volunteers will be asked to take off their shoes and weigh in light clothes.

Kinesio taping applications:

Two different kinesio taping applications will be applied to the patients by Dr. Figen Dağ. For both groups, first of all, the skin will be thoroughly cleaned of oil and moisture by means of alcohol cotton. As a result of the randomization, the group in which the 34 people to be included in the study was made from the web site (www.randomizer.org) . Patients will be blinded to the kinesio taping methods they will receive.

Pain and Ultrasonographic Evaluation:

Just before the kinesio taping application and immediately after the kinesio taping application (after 48 hours) after the bands are removed, the pressure pain assessment and the condition of the structures at the wrist level are blinded to the taping applications. It will be evaluated by Dr. Orhan GÜVENER (MD) by ultrasonography (US).

Pressure pain assessment will be carried out through a carpal tunnel with a mechanical algometer (J Tech Medical, Salt Lake City, UT, USA).

US measurements are carried out bidirectionally with linear probes (5-13 MHz Logiq P5; GE Medical Systems). Carpal tunnel evaluations will be performed while patients are seated with their hands in a neutral position. By avoiding compression of the probe on the tissue by using abundant gel, skin-subcutaneous tissue thickness, vertical, horizontal axle length and diameter of the median nerve, carpal ligament thickness, distance of carpal ligament and median nerve to the skin will be measured from proximal and distal carpal tunnel levels.

Presentation of Results and Statistical Methods to be used in the Study:

Statistical analyses will be made in a computer environment. The suitability of the variables to the normal distribution will be examined using visual (histogram and probability graphs) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). Demographic data, the results of the parameters to be evaluated will be evaluated by descriptive analyzes and will be given as mean (Average) ±standard deviation (SD), median, and/or interval. In the evaluation of intra-group differences, the paired-t-test will be used if the data show the normal distribution and Wilcoxon tests will be used if they do not show normal distribution. The differences between the groups will be determined by the independent t-test if the normal distribution of the data stops and by the Mann-Whitney U test if the normal distribution is not stopped. The relationships between the parameters will be examined using the Pearson test. For statistical analyses, the significance level will be considered to be 0.05.

Intergroup, 1st, and 2nd According to Cohen, at least 34 people were planned to be enrolled in the study to determine the significant difference between the measurements with 80% power and 5% type I error at 0.5 (moderate) effect size. The calculation was done in G*Power 3.1.9.4.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of moderate-mild carpal tunnel syndrome according to EMG findings
* Patients who read the informed consent form and volunteered to participate in the study

Exclusion Criteria:

* Patients with predisposing etiological factors (diabetes mellitus, acute trauma, rheumatological diseases, chronic kidney failure, pregnancy, hypothyroidism, hyperthyroidism, etc.) for carpal tunnel syndrome that may cause polyneuropathy.
* Patients receiving regular medical treatment such as continuous NSAIDs
* Patients who have received physical therapy or local steroid injection to the carpal tunnel region in the last 3 months
* Patients undergoing carpal tunnel surgery
* Patients with severe carpal tunnel syndrome
* Patients with a history of malignancy
* Patients with a history of cervical radiculopathy and ulnar neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Baseline ultrasonographic measurements | Just before Kinesio Taping application
  Ultrasonographic measurements will be made using linear probes (5-13 MHz Logiq P5; GE Medical Systems). Carpal tunnel assessments will be performed while the patients are sitting with their hands in a neutral position. By avoiding compression of the probe on the tissue by using plenty of gel, skin-subcutaneous tissue thickness, vertical and horizontal axis length and diameter of the median nerve, carpal ligament thickness, carpal ligament and median nerve distances to the skin will have measured. It will have measured in proximal and distal carpal tunnel levels.
After the application of ultrasonographic measurements | Immediately after the tapes are removed after the Kinesio Taping application (48 hours later)
  Ultrasonographic measurements will be made using linear probes (5-13 MHz Logiq P5; GE Medical Systems). Carpal tunnel assessments will be performed while the patients are sitting with their hands in a neutral position. By avoiding compression of the probe on the tissue by using plenty of gel, skin-subcutaneous tissue thickness, vertical and horizontal axis length and diameter of the median nerve, carpal ligament thickness, carpal ligament and median nerve distances to the skin will be measured from the proximal and distal carpal tunnel levels.
Baseline pain pressure threshold | Just before Kinesio Taping application
  Pain pressure threshold will be assessed through the carpal tunnel with a mechanical algometer (J Tech Medical, Salt Lake City, UT, USA).Assessments will be performed while the patients are sitting with their hands in a neutral position.
After the application of pain pressure threshold | Immediately after the tapes are removed after the Kinesio Taping application (48 hours later)
  Pain pressure threshold will be assessed through the carpal tunnel with a mechanical algometer (J Tech Medical, Salt Lake City, UT, USA).Assessments will be performed while the patients are sitting with their hands in a neutral position.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Güvener, MD, Principal Investigator — Mersin University Medical School; Figen Dağ, PhD, Study Chair — Mersin University
Locations (1):
- Mersin University Department of Physical Medicine and Rehabilitation, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guvener O, Dag F, Sahin G, Ozcakar L. Immediate effects of Kinesio taping in carpal tunnel syndrome: A randomized controlled double-blind ultrasonographic study. J Hand Ther. 2024 Oct-Dec;37(4):520-528. doi: 10.1016/j.jht.2023.12.017. Epub 2024 Feb 15. PMID 38360485